CLINICAL TRIAL: NCT07252297
Title: The Role of SIX6 as a Universal Cancer Marker in the Diagnosis of Non-Muscle Invasive Bladder Cancer
Brief Title: The Role of Universal Cancer Only Marker SIX6 in Diagnosing Non-Muscle Invasive Bladder Cancer
Acronym: NMIBC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XJLL-KY-20252509; 2024JC-YBQN-0984 (Other Grant/Funding Number: Shaanxi Province Natural Science Basic Research Program)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: DNA methylation;; biomarker; diagnosis
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: This study employs a parallel group design comparing two naturally occurring cohorts defined by SIX6 methylation status (positive vs. negative) in low-risk NMIBC patients, with prospective follow-up for recurrence outcomes.
Masking Description: This is a biomarker-based diagnostic study where participant grouping is determined by objective laboratory testing (SIX6 methylation status). Blinding of participants or investigators is not feasible due to the nature of the diagnostic assay.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIX6 Positive (Experimental): Participants with low-risk NMIBC who test positive for SIX6 gene methylation in their post-operative tissue or urine sample. This cohort is observed prospectively for the outcome of tumor recurrence.
  Interventions: Diagnostic Test: SIX6 Gene Methylation Assay
- SIX6 Methylation Negative (Experimental): Participants with low-risk NMIBC who test negative for SIX6 gene methylation in their post-operative tissue or urine sample. This cohort serves as the control and is observed prospectively for the outcome of tumor recurrence.
  Interventions: Diagnostic Test: SIX6 Gene Methylation Assay

INTERVENTIONS:
Diagnostic Test: SIX6 Gene Methylation Assay — A molecular diagnostic test that detects the methylation status of the SIX6 gene promoter region in post-operative tissue or urine samples from patients with low-risk non-muscle-invasive bladder cancer (NMIBC). The test uses quantitative methylation-specific PCR to determine methylation levels, which are then used to classify patients into SIX6 methylation positive or negative groups for prognostic assessment of recurrence risk.

SUMMARY:
Transurethral resection of bladder tumor (TURBT) is the standard therapeutic approach for patients with non-muscle-invasive bladder cancer (NMIBC). Postoperative intravesical chemotherapy or BCG immunotherapy is commonly administered to prevent recurrence. However, limitations such as suboptimal specimen integrity and tissue artifacts from intraoperative cauterization may lead to inaccurate risk stratification in cases classified as low-risk NMIBC, complicating individualized prognostic assessment. Consequently, clinicians often resort to prolonged intravesical therapy to mitigate recurrence risk, resulting in substantial overtreatment.

Previous studies in bladder cancer have demonstrated that detection of SIX6 gene methylation in urine enables noninvasive and accurate auxiliary diagnosis, with a sensitivity of 88.9%, specificity of 94.7%, and overall accuracy of 92.9%. In this retrospective case-control study, we aim to evaluate the utility of SIX6 methylation as an objective biomarker for predicting recurrence in patients with low-risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

1. age higher than 18;
2. patients diagnosis with non muscle invisive bladder cancer;
3. willing to provide 100Ml urine before treatment;
4. patients were diagnosis with bladder cancer for the first time

Exclusion Criteria:

1. patiens have more than one tumors besides bladder cancer;
2. pregnant women;
3. unwilling to partipate the research -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in SIX6 methylation levels between recurrence and non-recurrence groups | At the time of initial TURBT surgery (baseline)
  SIX6 gene promoter methylation level is measured as a continuous variable from post-operative tissue or urine DNA using quantitative methylation-specific PCR (qMSP). The values will be compared between the group of patients who later experience recurrence and the group who do not.

SECONDARY OUTCOMES:
Diagnostic performance of SIX6 methylation for predicting recurrence | Through study completion, up to 3 years
  The predictive performance will be assessed by calculating the Sensitivity, Specificity, Positive Predictive Value (PPV), Negative Predictive Value (NPV), and the Area Under the Receiver Operating Characteristic Curve (AUC-ROC) for the primary outcome of histologically confirmed tumor recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Xi Jing Hopspital, Xi'an, ShannxI, China

IPD SHARING:
Plan to Share IPD: No